CLINICAL TRIAL: NCT06400680
Title: Development of New Multifactorial Functional Evaluation Protocols and Related Indices for the Pediatric Age - Gait Spine Evaluation Protocol
Brief Title: Gait Spine Functional Evaluation Protocol
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1053
Record Dates: First submitted 2024-03-19; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Spine Disease; Gait
Keywords: Spine Kinematics; Thoracic Spine; Lumbar Spine; Motion analysis
MeSH Terms: conditions — Spinal Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy subjects (Experimental): Subjects without spine disease
  Interventions: Device: Spine Kinematic Assessment with Optoelectronic system
- Scoliotic subjects (Experimental): Subjects with a scoliosis diagnosis
  Interventions: Device: Spine Kinematic Assessment with Optoelectronic system

INTERVENTIONS:
Device: Spine Kinematic Assessment with Optoelectronic system — All measurements will be obtained using an optoelectronic multicamera system for human motion analysis (with eight high-resolution cameras with infrared light and a sampling frequency of 100 Hz.
  The experimental protocol require the positioning of markers (plastic spheres covered by reflecting film). Markers will be placed by clinical operators (physiotherapists with training in optoelectronic system for human motion analysis) after training and experience in recognition of the position of spinous and transversal processes, by manual identification.
  During the data acquisition protocol, the subject perform five trial of walking barefoot on a 6 m distance at a self-selected normal-pace speed.
  Every subject repeated this operations 2 times with 2 different operators.

SUMMARY:
The goal of this clinical trial is to develop and validate of a new protocol for multifactorial functional assessment of the kinematics of spinal and total body movements during walking by means of the optoelectronic motion analysis system in healthy and scoliosis subjects.

The main questions it aims to answer are:

* Is feasibility developing a protocol to assess the spine kinematic during walking?
* Is the intra and inter operator reliability of the developed protocol acceptable?
* Is the usability of the developed protocol acceptable? During data acquisition a trained therapist placed reflective markers on the skin of the participants in the selected body landmarks. The participants will be asked to perform five trial of walking barefoot on a 6 meters distance at a self-selected normal-pace speed, for each session.

DETAILED DESCRIPTION:
The spine is the central supporting structure of the body and for the torso in particular, allowing for flexibility and shock absorption, as well as routing and protecting the spinal cord and supporting the head and upper limbs for sensory and motor functions. In this perspective the evaluation of its movements in a global and segmental contribution is of paramount importance and cannot be separated by the other tasks. The locomotor function was the first one targeted by human motion analysis and still represent the main application in the rehabilitation. Optoelectronic systems are the gold standard technique for this assessment and specific protocols are available and applied. Traditional stereophotogrammetric models were used to assess the kinematics of pelvis, hip, knee, ankle, trunk (considered as a single rigid segment that does not provide information on kinematic changes within the spine). Indeed, it is relevant to understand the integrated and synergic motion of the spine and other body segment for a variety of applications, such as clinical diagnosis, endoprosthesis design, and the evaluation of treatment outcomes. Therefore, an accurate trunk motion analysis may be useful during medical diagnostic-therapeutic process. The aim of this study is introducing a new protocol consisting of a marker set, i.e. an innovative and integrated biomechanical model of the human body for the global analysis of spine and body movement during gait allows for a more detailed evaluation of the motor behavior and its abnormalities to better characterize the functionality of the spine at the level of its three main segments (upper thoracic, lower thoracic and lumbar), both on the sagittal, frontal and transversal plane, during walking. The development of a new protocol of analysis requires the validation before its definitive and clinical application. More in detail, the validation should be carried out in terms of both comparisons with reference absolute measures and the evaluation of its repeatability with healthy subjects.

ELIGIBILITY:
For healthy group:

Inclusion Criteria:

* no history of low back pain or spine related pathology

Exclusion Criteria:

* motor impairments during gait

For scoliosis group:

Inclusion Criteria:

* Diagnosis of idiopathic scoliosis
* Autonomous gait

Exclusion Criteria:

* motor impairments during gait

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-18 (Actual); Primary Completion 2026-05-18 (Estimated); Study Completion 2026-05-18 (Estimated)

PRIMARY OUTCOMES:
Intra/Inter Operator Reliability | Through study completion, an average of 3 year
  In the intra and interoperator repeatability analysis the investigators considered the correlation coefficient for the average RoM (in the 5 trials) in corresponding sessions. In particular, the investigators referred to standard interpretation criteria: the ICC values 0.5 and 0.75 indicate moderate reliability, values between 0.75 and 0.9 indicate good reliability, and values greater than, 0.90 indicate excellent reliability.
  Intra and inter operator reliability will be calculated at the achievement of ten healthy subjects ( during the first year), and then at the achievement of ten scoliotic subjects (during the second year)
Root mean square error as measure of accuracy | Year 1
  For the accuracy analysis, the comparison between the reference measures and the measure obtained with the optoelectronic system for every segment of the spine assessed through the root mean square error
SUS questionnaire score for usability assessment | Through study completion, an average of 3 year
  About the usability assessment, the System Usability Scale (SUS) collected at the end of each acquisition and calculated the average score value. The SUS provides a reliable tool for measuring the usability. The SUS questionnaire consists of a 10 item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Andreoni, Principal Investigator — IRCCS E. Medea - La Nostra Famiglia
Locations (1):
- IRCCS E. Medea, Bosisio Parini, Lecco, Italy